CLINICAL TRIAL: NCT03666910
Title: Assessment of Hearing in Children Born to Rheumatic Diseased Women Treated With Antimalarial Drugs During Pregnancy
Brief Title: Hearing Problems in Children of Rheumatic Diseased Mothers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Ragab Mohasseb Ali, Principle investigator, Assiut University
Other Study IDs: 17100500
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Hearing Disorders
MeSH Terms: conditions — Hearing Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- children of rheumatic diseased mothers not on treatment
  Interventions: Diagnostic Test: Audiometer
- children of rheumatic diseased mothers on antimalarial drugs
  Interventions: Diagnostic Test: Audiometer
- children of normal mothers
  Interventions: Diagnostic Test: Audiometer

INTERVENTIONS:
Diagnostic Test: Audiometer — detection of hearing problems

SUMMARY:
Evaluation of the hearing functions of children born to rheumatic diseased mothers who received gestational antimalarial drugs versus those didn't receive gestational antimalarials drugs compared with normal healthy children.

DETAILED DESCRIPTION:
Rheumatic diseases are autoimmune illnesses characterized by tissue damage, caused by abnormal immunologic reaction against own cells, tissues or organs.Many of these rheumatic diseases preferentially occur in women during the childbearing age.

The transplacental passage of maternal antibody may result in a variety of adverse fetal effects including thrombocytopenia, neutropenia, hemolysis and thyroid disease. Both fetal hypo and hyper thyroidism may occur and maternal hypothyroidism particularly during the 1st trimester is associated with impaired fetal neurological development and delayed mental and motor development.

Hydroxychloroquine (CQ), the hydroxyl derivative of chloroquine, is an antimalarial agent which is widely used, either alone or in combination with other agents, in the treatment of SLE, rheumatoid arthritis (RA) and various other autoimmune diseases.

Hydroxychloroquine is safe during pregnancy, as it is not associated with an increased rate of congenital malformations. However, isolated cases of ocular (retinal pigment deposits) and auditory abnormalities were reported.

An increase in high-frequency hearing threshold is the earliest change in the auditory function for most drug induced hearing losses, including the irreversible damage caused by antimalarials.

The investigators therefore will use audiological methods for detection of hearing impairment in children delivered for mothers receiving antimalarials during pregnancy with rheumatic diseases.

ELIGIBILITY:
Inclusion Criteria:

* children males & females
* Age 4 to 16 years.
* whose mothers have rheumatic diseases during pregnancy with gestational intake of antimalarial drugs as a treatment.

Exclusion Criteria:

* Prematurity, history of prenatal, natal or post natal medical problems.
* Family history +ve.
* Consanguinity +ve.
* Gestational intake of other ototoxic drugs.
* Use of antimalarial due to diseases other than rheumatic diseases.
* Administration of antimalarial before pregnancy.
* Children who have middle ear disorders.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children (age 4 to 16 years) whose mothers have rheumatic diseases during pregnancy with gestational intake of antimalarial drugs as a treatment.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Dual channel audiometer | 20 mimutes
  evaluate the hearing functions of children born to rheumatic diseased mothers who received gestational antimalarial drugs versus those didn't receive gestational antimalarials drugs compared with normal healthy children.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Ragab mohasseb, Phd, Principal Investigator — Assiut University

REFERENCES:
- [Background] Baldwin C, Avina-Zubieta A, Rai SK, Carruthers E, De Vera MA. Disease-modifying anti-rheumatic drug use in pregnant women with rheumatic diseases: a systematic review of the risk of congenital malformations. Clin Exp Rheumatol. 2016 Mar-Apr;34(2):172-83. Epub 2016 Mar 3. PMID 26940667